CLINICAL TRIAL: NCT05584332
Title: A Multicenter,Randomized, Placebo-Controlled, and Double-blind Phase Ⅲ Study to Evaluate the Efficacy, Immunogenicity and Safety of Quadrivalent Human Papillomavirus (Types 6, 11, 16, and 18) Recombinant Vaccine (Hansenula Polymorpha) in Chinese Female Aged 18-45 Years
Brief Title: A Phase Ⅲ Study to Evaluate the Efficacy, Immunogenicity, Safety of Quadrivalent HPV Recombinant Vaccine in Chinese Healthy Females
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Strategic adjustment
Sponsor: Shanghai Bovax Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4-HPV-3004
Record Dates: First submitted 2022-10-12; First posted 2022-10-18 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2022-10

CONDITIONS: Cervical Cancer; Genital Wart; CIN1; CIN2; CIN3; Vain I; Vain III; Vin I; Vin II; Vin III; AIS; VAIN - Vaginal Intraepithelial Neoplasia 2
MeSH Terms: conditions — Uterine Cervical Neoplasms; Condylomata Acuminata | interventions — Vaccines, Synthetic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo
- 4vHPV Vaccine (Experimental)
  Interventions: Biological: Quadrivalent Human Papillomavirus (Types 6, 11, 16, and 18) Recombinant Vaccine (Hansenula Polymorpha)

INTERVENTIONS:
Biological: Quadrivalent Human Papillomavirus (Types 6, 11, 16, and 18) Recombinant Vaccine (Hansenula Polymorpha) — 0.5 ml injection in 3 dosing regimen
  Arms: 4vHPV Vaccine
Biological: Placebo — 0.5 ml injection in 3 dosing regimen
  Arms: Placebo

SUMMARY:
This study is designed to evaluate the vaccine efficacy, immunogenicity and safety of the 4-valent Human Papillomavirus (Types 6, 11, 16, and 18) Recombinant Vaccine (Hansenula Polymorpha) in Chinese Female Subjects Aged 18-45 Years .

ELIGIBILITY:
Inclusion Criteria:

* (IF Non-compliance with criterion "*" option, the visit WILL be rescheduled)

  1. Chinese women aged 18-45 who can provide legal identification and had a sexual life history;
  2. The subject fully understands the study procedures, understands the risks and benefits associated related this study, and voluntarily signs the informed consent;
  3. Subjects are able to read, understand and fill in application forms such as diary CARDS and contact CARDS, and participate in regular follow-up visits according to the study protocol;
  4. *axillary's temperature <37.3℃ on the day of enrollment;
  5. Subjects have not received any form of cervical cancer screening, or have been received but the results are normal;
  6. *0 days before the gynecological visit, no sex within 48 hours, no flushing or vaginal cleaning within 72 hours, no use of vaginal drugs or preparations;
  7. When the subjects were enrolled, the urine pregnancy test was negative (sensitivity was 25mIU/ml β-HCG), they were not in the lactation period, had no family planning from Day 0 to 30 days after receiving the third dose of the vaccine. Agree to continue to use effective contraception (including: oral contraceptives, injectable or embedded contraceptives, sustained-release topical contraceptives, hormone patches, intrauterine devices (IUDs), sterilization, abstinence, condoms (men), diaphragms, cervical caps, etc.) from the day of enrollment to 30 days after the third season of vaccination. Safe-period contraception, in vitro ejaculation, and emergency contraception are unacceptable methods of contraception.

Exclusion Criteria:

* (IF Non-compliance with criterion "*" option, the visit WILL be rescheduled)

  1. Blood pressure (BP) before the first dose of vaccination was higher than normal or increased (systolic BP ≥140mmHg and/or diastolic BP ≥90mmHg);
  2. * Subjects had fever symptoms (axillary's temperature ≥37.3℃) before the first day of vaccination (within 24 hours before vaccination);
  3. History of severe side effect to previous vaccinations or History of severe allergies (e.g. Swelling of the mouth and throat, Dyspnea, Hypotension or Shock, Severe urticaria) to components of study vaccine (e.g. Histidine, Polysorbate, and Aluminium phosphate). History of severe allergies requiring medical intervention, such as anaphylactic shock, anaphylactic laryngeal edema, allergic purpura, thrombocytopenic purpura, local allergic necrosis reaction (Arthus reaction), etc;
  4. Subjects with compromised immune systemsor have been diagnosed with congenital or acquired immune deficiency, HIV infection, lymphoma, leukemia, systemic lupus erythematosus (SLE), rheumatoid arthritis, juvenile rheumatoid arthritis (JRA), inflammatory bowel disease or Autoimmune thyroid disease （e.g. Hyperthyroidism，Thyroiditis/Subacute thyroiditis，or Hypothyroidism), and other Autoimmune diseases ;
  5. Previous or current have epilepsy, seizures (except febrile seizures in children) or convulsions, or mental diseases, with a family history of psychosis;
  6. Absence of spleen or functional absence of spleen, and absence of spleen or splenectomy in any case;
  7. Previous or current have severe liver, kidney and cardiovascular diseases, diabetic complications or malignant tumor;
  8. Patients with thrombocytopenia or any coagulation disorders that may be contraindications to intramuscular injection;
  9. Immunosuppressant or immunopotentiator therapy within 1 month before the first dose of vaccination, such as long-term use of systemic glucocorticoid therapy (≥2mg/kg/ day, for more than 2 weeks, such as prednisone or similar drugs;Topical administration (such as ointment, eye drops, inhalant or nasal spray) exceeding the recommended dosage in the directions or showing any signs of systemic exposure) or planning to receive such treatment between the day of the first dose and 30 days after the third dose of the vaccine;
  10. Received any immunoglobulin or blood product within 3 months prior to the first dose of vaccination, or plans to receive such product between the day of the first dose and 30 days after the third dose of the vaccine;
  11. * An acute illness or an acute episode of a chronic illness within 3 days prior to vaccination, or use antipyretic, analgesic and antiallergic drugs (e.g., acetaminophen, ibuprofen, aspirin, loratadine, cetirizine, etc.);
  12. Have participated in other gynecology-related clinical trials within 6 months, and have used or plan to use other investigational or unregistered products (drugs or vaccines) other than the vaccine in this study within 3 months;
  13. * Received inactivated/recombinant/DNA vaccines (Non-attenuated vaccines) within 14 days prior to enrollment, or attenuated live vaccines within 28 days prior to enrollment;
  14. Have been vaccinated with commercially available HPV vaccine in the past or planned to be vaccinated with commercially available HPV vaccine during the study period;Or have participated in a clinical trial of the HPV vaccine and have received a vaccine/placebo vaccination;
  15. Subjects may be unable to comply with the study procedure, comply with the agreement, or plan to permanently relocate from the region prior to completion of the study, or may be permanently absent from the region during the scheduled visit;
  16. In the opinion of the investigators, the subjects had any other factors that made them unsuitable to participate in the clinical trial, so that continued participation in the study could not guarantee the maximum benefit of the subjects;
  17. * The first dose of vaccine was in pregnancy at the time of vaccination, or the end of pregnancy had not exceeded 6 weeks;
  18. * Subject is in the menstrual period;
  19. Previous positive history of HPV;
  20. Had a history of abnormal cervical cytology, including squamous intraepithelial lesions (SIL) or not clear meaning of the atypical squamous cells (ASC - US), except the atypical squamous cells - not highly squamous intraepithelial lesion (ASC - H), atypical glandular epithelial cells, or those with cervical intraepithelial neoplasia (CIN) and carcinoma in situ or abnormal cervical biopsy results such as the history;
  21. Previous history of vulvar intraepithelial neoplasia, vaginal intraepithelial neoplasia, genital warts, vulvar cancer, vaginal cancer, cancer, etc. may be caused by HPV infection;
  22. Received total hysterectomy or pelvic radiotherapy;
  23. Cervical insufficiency or abnormal cervical structure (judged by the results of routine gynecological examination);
  24. Previous sexual history (including syphilis, gonorrhea, chancre, venereal lymphatic granuloma, granuloma inguinal) or had a history of condyloma;
  25. Gynecological examination before the first dose of vaccination suspected genital warts, or on the basis of clinical symptoms and signs suspected vulva, vagina or cervical precancerous lesions and the possibility of cancer.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3131 (Actual)
Dates: Start 2022-12-09 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-23 (Actual)

PRIMARY OUTCOMES:
The person-year incidence of HPV 16 and 18-related CIN 2+ observed in Chinese women aged 18-45 years after receiving 3 doses of quadrivalent HPV vaccine at least 30 days ago. | Over 30 months

SECONDARY OUTCOMES:
The person-year incidence of HPV 6-, 11-, 16-, and 18-related 6-month Persistent Infection at least 30 days post Dose 3 | from Month 7 up to Month 60
The person-year incidence of HPV 6-, 11-, 16-, and 18-related 12-month Persistent Infection at least 30 days post Dose 3 | from Month 7 up to Month 60
The person-year incidence of HPV 6-, 11-, 16-, and 18-related disease (e.g., VIN1+ orAIN1+ or VAIN1+ and genital warts) | from Month 7 up to Month 60
Percentage of Participants Who Report at any Injection-site and Systemic Adverse Event 30 minutes post any vaccination | 30 minutes after any dose of vaccination
Number of subjects with Adverse Events (AEs) | From Day 0 to Month 30
  Subjects with solicited and unsolicited AEs
Number of subjects with Severe adverse events (SAE) | Through study completion，expected 60 months
  SAEs assessed include medical occurrences that results in death, are life threatening, require hospitalization or prolongation of hospitalization, results in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subjects.
Number of subjects with pregnancy events | Through study completion，expected 60 months
  Outcomes of pregnancies were Live infant NO apparent congenital anomaly (ACA) , Live infant, Elective termination NO ACA, Elective termination CA, Ectopic pregnancy, Spontaneous abortion NO ACA, Stillbirth, Lost to follow up and Pregnancy ongoing.
Number of subjects receiving the whole schedule vaccination with antibody responses as assessed by SCR | Month7
The neutralizing antibody level among the subjects receiving the whole schedule vaccination | Month7
The person-year incidence of non-vaccine-realted HPV types related CIN2+ observed in Chinese women aged 18-45 years at least 30 days post Dose 3 | Through study completion，expected 60 months
The person-year incidence of non-vaccine-realted HPV types related disease (e.g., VIN1+ or AIN1+ or VAIN1+ and genital warts) observed in Chinese women aged 18-45 years at least 30 days post Dose 3 | Through study completion，expected 60 months
The person-year incidence of HPV 6-, 11-, 16-, and 18-related 6-month and 12-month Persistent Infection at least 30 days post Dose 1 | From Month 1 up to Month 60
The person-year incidence of HPV 16- and 18-related CIN2+ at least 30 days post Dose 1 | From Month 1 up to Month 60
The person-year incidence of HPV 6-, 11-, 16- and 18-related diseases (e.g., VIN1+ or AIN1+ or VAIN1+ and genital warts) at least 30 days post Dose 1 | From Month 1 up to Month 60

CONTACTS AND LOCATIONS:
Locations (1):
- Yi M, Liuchow, Guangxi, China